CLINICAL TRIAL: NCT01882634
Title: Screening Programme for Abdominal Aortic Aneurysm by Hand-Held-Ultrasonography in Primary Health Care
Acronym: BarcelonAAA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Consorci d'Atenció Primària de Salut de l'Eixample (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Antoni Siso Almirall, Head of Research, Consorci d'Atenció Primària de Salut de l'Eixample
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CP041192
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound arm (Experimental)
  Interventions: Device: Ultrasound (Trademark:VScan; Manufacturer:General Electric)

INTERVENTIONS:
Device: Ultrasound (Trademark:VScan; Manufacturer:General Electric) — Standardized measurements were made and aorta will be visualized in a minimum of three hard copy images: upper transverse projection abdominal aorta at the level of epigastrium (celiac trunk) lower transverse section for distal view of aorta (pre-bifurcation), and longitudinal section (with origin of celiac trunk or superior mesenteric artery), determining the maximum diameter in centimeters (cm)

SUMMARY:
To determine the prevalence of Abdominal Aortic Aneurysm (AAA) in the Spanish men over 60 years through a screening program in Primary Health Care using a hand-held ultrasound and to analyze the relationship between cardiovascular risk factors and cardiovascular disease in patients with AAA.

DETAILED DESCRIPTION:
Study includes a cohort of men over 60 years attented in primary health care centers of Consorci d'Atenció Primària de Salut d'Eixample (CAPSE).General practitioners complete an ultrasonography training in an ultrasound unit under supervision of experienced radiologists using a standard ultrasound equipment and hand-held ultrasound (Trademark: VScan, Manufacturer: General Electric, USA). All images and video are blindly evaluated by a radiologist in order to establish the concordance in the interpretation of images between general practitioners and radiologist. Kappa index will be used to study the agreement on the presence or absence of AAA. Multivariate logistic regression analysis will be used to determine the factors that influence the presence of AAA.

ELIGIBILITY:
Inclusion Criteria:

* Men 60 years or more
* Attending at primary health care center for any complaint

Exclusion Criteria:

* Subjects being hemodynamically unstable at presentation
* Subjects with previous AAA confirmed by abdominal ultrasound scan or another image diagnosis technique
* Subjects deemed to require emergent treatment at presentation or after initial history and physical examination.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The prevalence of abdominal aortic aneurysm detected by a hand-held ultrasound in Primary Care | 12 months

SECONDARY OUTCOMES:
Associated risk factors to abdominal aortic aneurysm | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Sisó Almirall, MD PhD, Principal Investigator — Head of Research - Consorci d'Atenció Primària de Salut Eixample (CAPSE); Daniel Cararach Salami, MD, Study Chair — General Practitioner. Primary Care Center Les Corts, Consorci d'Atenció Primària de Salut Eixample (CAPSE); Alfonso Pérez Jiménez, MD, Study Chair — General Practitioner. Primary Care Center Casanova, Consorci d'Atenció Primària de Salut Eixample (CAPSE); Marta Navarro González, MD, Study Chair — General Practitioner. Primary Care Center Comte Borrell, Consorci d'Atenció Primària de Salut Eixample (CAPSE); Rosa Gilabert Solé, MD PhD, Study Chair — Radiologist. Senior Consultant. Department of Radiology, Hospital Clínic; Concepció Bru Saumell, MD PhD, Study Chair — Radiologist. Senior Consultant. Department of Radiology, Hospital Clínic; Vicenç Riambau Alonso, MD PhD, Study Chair — Chief of Vascular Surgery Division, Thorax Institute, Hospital Clinic; Laura Sebastián Montal, MD, Study Chair — General Manager in Consorci d'Atenció Primària de Salut Eixample (CAPSE); Jaume Benavent Àreu, MD, Study Chair — Director d'Afers Assistencials. Catalan Institute of Health. Ministry of Health. Catalonia, Spain.; Belchin Kostov, MSc, Study Chair — Statistician. Transverse Group for Research in Primary Care, IDIBAPS.
Locations (3):
- Spain (3):
  - Primary Care Center Les Corts, Barcelona, Catalonia
  - Primary Care Center Casanova, Barcelona, Catalonia
  - Primary Care Center Comte Borrell, Barcelona, Catalonia